CLINICAL TRIAL: NCT06802952
Title: RTMS for Clinical High-risk Syndrome of Psychosis Based on Personalized Targets Using Magnetoencephalography
Brief Title: RTMS for CHR Based on Personalized Targets Using Magnetoencephalography
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MEG-CHR-2024
Record Dates: First submitted 2025-01-26; First posted 2025-01-31 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-01

CONDITIONS: Clinical High-risk Syndrome of Psychosis
Keywords: Clinical high-risk syndrome of psychosis; MEG; rTMS; Individualized targets

STUDY DESIGN:
Intervention Model Description: Exploratory self controlled clinical intervention trial. Pseudo stimulus intervention in weeks 1-2, for a total of 10 days. After resting for 2 weeks, enter the 3-4 weeks of real stimulation, with 5 days of intervention per week for a total of 10 days.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Physical intervention for before-after study in the same subject with CHR (Other): Pseudo stimulus intervention in weeks 1-2, for a total of 10 days. After resting for 2 weeks, enter the 3-4 weeks of real stimulation, with 5 days of intervention per week for a total of 10 days.
  Interventions: Device: rTMS

INTERVENTIONS:
Device: rTMS — RTMS using pseudo stimulus intervention in weeks 1-2, for a total of 10 days. After resting for 2 weeks, enter the 3-4 weeks of real stimulation, with 5 days of intervention per week for a total of 10 days. Application of rTMS for 1Hz low-frequency intervention, with intervention parameters of 1400 sessions, 100% exercise threshold, and a total of 23 minutes per session. After each target intervention, rest for half an hour to one hour.

SUMMARY:
This study is an before-after study in the same subject, which enrolled 26 individuals with high-risk psychiatric syndrome (CHR). The target of subjects intervention relies on the results of magnetoencephalography localization. The medication and dosage remain unchanged during the intervention period or not yet taking antipsychotic medication. The investigators assume that the intervention targets for each CHR subject are individualized.

DETAILED DESCRIPTION:
This study is divided into two parts:

1. Target determination. Firstly, MEG data of the subject's resting and task states are collected, and a precise localization model using magnetoencephalography is applied to locate the precise location of the subject's abnormal signals in the brain, which is then used as the intervention target. Based on the subject's tolerance for single day intervention, the appropriate number of targets is generally 2-4. The upper limit of targets is 4.
2. RTMS individualized intervention. Application of rTMS for 1Hz low-frequency intervention, with intervention parameters of 1400 sessions, 100% exercise threshold, and a total of 23 minutes per session. After each target intervention, rest for half an hour to one hour. The pseudo stimulation intervention lasted for 10 days in the first and second weeks, and the scale was evaluated after the end of the pseudo stimulation. After resting for 2 weeks, enter the 3-4 weeks of real stimulation, with 5 days of intervention per week for a total of 10 days. 2-4 targets per day, 23 minutes per target, with 30-60 minutes between interventions for each target. After the fourth week, evaluate the scale. Follow up evaluations will be conducted on the 7th, 14th, 30th, 60th, and 90th day after intervention. By analyzing and evaluating data, explore individualized treatment plans for CHR in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Clinical High-Risk Syndrome for Psychosis
* Must be able to right-handed
* Primary school education or above
* Understand and sign a written informed consent form (jointly signed by the guardian and the participant if under 18 years old)

Exclusion Criteria:

* Major physical illnesses (organic lesions such as sensory and motor disorders, neurological disorders, and traumatic brain injury)
* Taboo symptoms for rTMS treatment (such as intracranial metal implants)
* Metal (including orthodontic treatment, dental implants) and tattoos inside the body
* Claustrophobia

Ages: 13 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-02-07 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Reduction rate of the SIPS/SOPS scale | From enrolment to the end of the 2-week pseudostimulation treatment. From 2 weeks rest after the end of pseudostimulation treatment to the end of 2 weeks of true stimulation treatment.
  SIPS/SOPS (Structured Interview for Psychosis-Risk Syndromes/Scale of Psychosis-Risk Symptoms) is a scale used to assess subjects' structural interviews on prodromal symptoms of psychosis. The SIPS/SOPS scales, due to their inclusion of multiple assessment items with potentially varying scores for each, do not allow for a straightforward determination of an overall minimum and maximum value. A higher score indicates more severe symptoms in the assessed individual, while a lower score suggests less severe symptoms.

SECONDARY OUTCOMES:
Reduction rate of the PNASS scale | From enrolment to the end of the 2-week pseudostimulation treatment. From 2 weeks rest after the end of pseudostimulation treatment to the end of 2 weeks of true stimulation treatment.
  PNASS (Positive and Negative Syndrome Scale) is a scale for evaluating Psychiatric disorders. Each item is scored on a scale from 1 to 7, with 1 being the lowest score and 7 being the highest. Therefore, the minimum possible score on the PANSS is 30, and the maximum is 210. A higher score indicates more severe symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Mental Health Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided
All research data sharing related to humans requires hospital approval.

REFERENCES:
- [Background] Tang Y, Xu L, Zhu T, Cui H, Qian Z, Kong G, Tang X, Wei Y, Zhang T, Hu Y, Sheng J, Wang J. Visuospatial Learning Selectively Enhanced by Personalized Transcranial Magnetic Stimulation over Parieto-Hippocampal Network among Patients at Clinical High-Risk for Psychosis. Schizophr Bull. 2023 Jul 4;49(4):923-932. doi: 10.1093/schbul/sbad015. PMID 36841956
- [Background] Zhang T, Xu L, Wei Y, Cui H, Tang X, Hu Y, Tang Y, Wang Z, Liu H, Chen T, Li C, Wang J. Advancements and Future Directions in Prevention Based on Evaluation for Individuals With Clinical High Risk of Psychosis: Insights From the SHARP Study. Schizophr Bull. 2025 Mar 14;51(2):343-351. doi: 10.1093/schbul/sbae066. PMID 38741342